CLINICAL TRIAL: NCT02799667
Title: Randomized Controlled Trial: Do Single Use Negative Pressure Dressings Reduce Wound Complications in Women With a BMI >40 kg/m2 Undergoing Cesarean Delivery at a Tertiary Medical Center?
Brief Title: Do Single Use Negative Pressure Dressings Reduce Wound Complications in Obese Women After Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11943
Record Dates: First submitted 2016-05-20; First posted 2016-06-15 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Surgical Site Infections; Wound Complications; Complications; Cesarean Section
Keywords: negative pressure wound therapy; cesarean delivery
MeSH Terms: conditions — Obesity; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dressing (Active Comparator): Women will be randomized to receive the standard dressing (sterile gauze, non absorbent sterile gauze, and a waterproof bandage) at the time of fascial closure in a cesarean delivery.
  Interventions: Device: Standard Dressing
- Negative Pressure Wound Therapy Dressing (Experimental): Women will be randomized to receive the Negative Pressure Wound Therapy (NPWT) dressing at the time of fascial closure in a cesarean delivery.
  Interventions: Device: Negative Pressure Wound Therapy Dressing

INTERVENTIONS:
Device: Standard Dressing — Patients are randomized to the standard dressing at the time of fascial closure.
  Arms: Standard Dressing
Device: Negative Pressure Wound Therapy Dressing — Patients are randomized to the NPWT at the time of fascial closure.
  Arms: Negative Pressure Wound Therapy Dressing

SUMMARY:
The investigators aim to show that single use negative pressure dressings can decrease the rate of wound complications in obese women (BMI > 40 kg/m2) undergoing cesarean delivery at a tertiary medical center by randomizing women to receive either a single use negative pressure dressing or the standard dressing after cesarean delivery.

DETAILED DESCRIPTION:
Subjects admitted to L+D for obstetric or medical indications at a tertiary medical center with a BMI > 40 kg/m2 will be asked to participate in a study on post surgical dressings and wound outcomes if they undergo cesarean delivery. Subjects will be randomized to either study arm at the time of fascial closure during cesarean delivery. Post operative care will not be altered. Incisions will be evaluated prior to hospital discharge. Subjects will present for a wound evaluation 2 weeks post operatively, and receive phone calls to assess outcomes at both 2 and 6 weeks post operatively.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 kg/m2 undergoing cesarean delivery for any cause and willing to have a 2 week post operative follow-up for a wound evaluation at Tufts Medical Center.

Exclusion Criteria:

* Women less than age 18, women with an active infection in the location of Pfannenstiel skin incision, women not willing to come to Tufts Medical Center for a wound evaluation 2 weeks post operatively, women who do not have height and weight information available, and women with a BMI < 40 kg/m2 will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael House, MD, Principal Investigator — Tufts Medical Center, physician
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterson AT, Bakaysa SL, Driscoll JM, Kalyanaraman R, House MD. Randomized controlled trial of single-use negative-pressure wound therapy dressings in morbidly obese patients undergoing cesarean delivery. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100410. doi: 10.1016/j.ajogmf.2021.100410. Epub 2021 May 28. PMID 34058423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Started | 55 | 55
Completed | 54 | 54
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 55 | 110
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (5.3) | 31.5 (6.3) | 31.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 14 | 22
  Not Hispanic or Latino | 47 | 41 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 38 | 41 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 55 | 110
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 47.8 (6.9) | 49.3 (6.6) | 48.6 (6.8)
gestational age [Mean (Standard Deviation); unit: weeks] | 36.4 (3.3) | 37.4 (3.1) | 36.9 (3.2)
gestational diabetes [Count of Participants; unit: Participants] | 20 | 15 | 35
pregestational diabetes [Count of Participants; unit: Participants] | 6 | 9 | 15
current smoker [Count of Participants; unit: Participants] | 2 | 4 | 6
former smoker [Count of Participants; unit: Participants] | 9 | 6 | 15
chronic steroid use [Count of Participants; unit: Participants] | 1 | 0 | 1
Insulin use [Count of Participants; unit: Participants] | 13 | 15 | 28
Oral Hypoglycemic agent use [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Outcome of the Presence of Wound Complications Diagnosed by the Two Week Post Operative Appointment
Description: Composite outcome of wound complications, defined as the presence of any of the following: superficial, deep, and organ space surgical site infections (SSIs), skin blisters around the incision, scar separation >1 cm, seroma requiring evacuation, hematoma requiring evacuation, wound debridement, hospital re-admission, and additional operating room management.
Time Frame: 2 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants | 14 | 10

2. Secondary Outcome: Number of Participants With Individual Wound Complications Diagnosed by the Two Week Post Operative Appointment
Description: The presence of each the following individual wound complications will be analyzed as separate outcomes: superficial, deep, and organ space SSIs, skin blisters around the incision, scar separation >1 cm, seroma requiring evacuation, hematoma requiring evacuation, wound debridement, hospital re-admission, and additional operating room management.
Time Frame: 2 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants
  superficial SSI: yes | 6 | 7
  superficial SSI: no | 49 | 48
  deep SSI: yes | 0 | 0
  deep SSI: no | 55 | 55
  organ space SSI: yes | 0 | 0
  organ space SSI: no | 55 | 55
  skin blisters: yes | 5 | 1
  skin blisters: no | 50 | 54
  scar separation: yes | 5 | 2
  scar separation: no | 50 | 53
  seroma w/evacuation: yes | 1 | 2
  seroma w/evacuation: no | 54 | 53
  hematoma w/evacuation: yes | 0 | 1
  hematoma w/evacuation: no | 55 | 54
  wound debridement: yes | 1 | 2
  wound debridement: no | 54 | 53
  hospital readmission: yes | 1 | 1
  hospital readmission: no | 54 | 54
  additional operative room management: yes | 0 | 1
  additional operative room management: no | 55 | 54

3. Secondary Outcome: Number of Participants With Composite Outcome of the Presence of Severe Wound Complications Diagnosed by the Two Week Post Operative Appointment
Description: Composite outcome of the presence of one of the following major complications; deep incisional SSIs, scar separation > 1 cm, seroma requiring evacuation, hematoma requiring evacuation, wound debridement, hospital readmission and additional operating room management.
Time Frame: 2 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants | 11 | 5

4. Secondary Outcome: Number of Participants With Composite Outcome of the Presence of Wound Complications Diagnosed at a Two Week Post Operative Appointment, or Ascertained Through Patient Phone Calls at 2 and 6 Weeks Post Operatively.
Description: as for outcome 1
Time Frame: 6 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants | 16 | 11

5. Secondary Outcome: Number of Participants With Individual Wound Complications Diagnosed at a Two Week Post Operative Appointment or Ascertained Via Patient Phone Calls at 2 and 6 Weeks Post Operatively
Description: as for outcome 2
Time Frame: 6 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants
  superficial SSI: yes | 7 | 7
  superficial SSI: no | 48 | 48
  deep SSI: yes | 0 | 0
  deep SSI: no | 55 | 55
  organ space SSI: yes | 0 | 0
  organ space SSI: no | 55 | 55
  skin blisters: yes | 5 | 2
  skin blisters: no | 50 | 53
  scar separation: yes | 7 | 2
  scar separation: no | 48 | 53
  seroma w/evacuation: yes | 1 | 2
  seroma w/evacuation: no | 54 | 53
  hematoma w/evacuation: yes | 0 | 1
  hematoma w/evacuation: no | 55 | 54
  wound debridement: yes | 1 | 2
  wound debridement: no | 54 | 53
  hospital readmission: yes | 1 | 1
  hospital readmission: no | 54 | 54
  additional operative room management: yes | 0 | 1
  additional operative room management: no | 55 | 54

6. Secondary Outcome: Number of Participants With Composite Outcome of the Presence of Severe Wound Complications Diagnosed at a Two Week Post Operative Appointment or Ascertained Via Patient Phone Calls at 2 and 6 Week Post Operatively
Description: as for outcome 3
Time Frame: 6 weeks post partum/post operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
Number analyzed (Participants) | 55 | 55
Participants | 12 | 5

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Standard Dressing | Negative Pressure Wound Therapy Dressing
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

LIMITATIONS AND CAVEATS:
Early termination secondary to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02799667/Prot_SAP_ICF_000.pdf